CLINICAL TRIAL: NCT05856448
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally Administered GLPG3667 in Adult Subjects With Active Systemic Lupus Erythematosus
Brief Title: A Study Evaluating the Effects of GLPG3667 Administered as Oral Treatment in Adult Participants With Active Systemic Lupus Erythematosus
Acronym: GALACELA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG3667-CL-215; 2023-503183-16-00 (EU CTIS Number)
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GLPG3667 - Treatment A (Experimental): Participant will receive a dose A of GLPG3667 capsules orally once daily (q.d.) for 48 weeks.
  Interventions: Drug: GLPG3667
- GLPG3667 - Treatment B (Experimental): Participant will receive a dose B of GLPG3667 capsules orally (q.d.) for 48 weeks.
  Interventions: Drug: GLPG3667
- Placebo (Placebo Comparator): Participant will receive placebo matched to GLPG3667 capsules orally q.d for 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG3667 — Capsule
  Arms: GLPG3667 - Treatment A; GLPG3667 - Treatment B
Drug: Placebo — Capsule
  Arms: Placebo

SUMMARY:
A study evaluating the efficacy, safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of GLPG3667 administered orally once daily for 48 weeks in approximately 180 adult participants with active Systemic Lupus Erythematosus (SLE).

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant with documented diagnosis of SLE as defined by the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria with a disease diagnosed ≥24 weeks before the screening visit.
2. Participant has a total Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥6 points and a clinical SLEDAI-2K score ≥4 at screening and baseline (scores must be confirmed by central review at screening).

   * Lupus headache, alopecia, organic brain syndrome, and mucous membrane ulceration will not count toward the score required for screening at entry.
   * Clinical SLEDAI-2K excludes laboratory abnormalities such as hematuria, pyuria, urinary casts, proteinuria, positive anti-double-stranded deoxyribonucleic acid (anti-dsDNA), decreased complement, thrombocytopenia, and leukopenia.
3. Participant is positive for 1 of the following: antinuclear antibodies (ANA) ≥1:80 or positive anti-dsDNA (indeterminate values are considered positive), or positive anti-Smith (anti-Sm), as determined by the central laboratory.
4. At least 1 of the following BILAG-based protocol-specific manifestations of SLE:

   * BILAG A or B score in the mucocutaneous body system.
   * BILAG A or B score in the musculoskeletal body system due to arthritis.
   * If only 1 B and no A score is present in the mucocutaneous body system or in the musculoskeletal body system due to arthritis, then at least 1 B score must be present in one of the other body systems, for a total of >=2 BILAG B body system scores.
5. Background therapy with at least 1 of the following medications is required for >=12 weeks before the screening visit and must remain stable until randomization and throughout study participation:

   * 1 immunosuppressant (combination of immunosuppressants is not permitted), stable at least 8 weeks prior to screening.
   * 1 antimalarial, stable at least 8 weeks prior to screening. In addition, oral corticosteroids (CS) (prednisone or equivalent) and/or NSAIDs background therapy is permitted but not required:
   * CS (prednisone or equivalent; <=30 mg/day; CS monotherapy is not permitted), stable at least 2 weeks prior to screening; AND/OR
   * Non-steroidal anti-inflammatory drugs (NSAIDs; NSAIDs monotherapy is not permitted), stable at least 2 weeks prior to screening.

Key Exclusion Criteria:

1. Participant with active, severe lupus nephritis (World Health Organization Class III, IV) that requires or may require treatment with cytotoxic agents or high-dose CS are excluded.
2. Participants with pre-existing, controlled renal disease with serum creatinine≥ 2 x upper limit of normal (ULN) and either residual proteinuria up to 3 grams/day (g/day) or a urine protein: creatinine ratio (UPCR) of up to 3 milligrams/milligrams (mg/mg) or 339 milligrams of albumin per millimole of creatinine (mg/mmol) are allowed. Control of renal disease must be documented with at least 2 measurements of proteinuria or UPCR over the past 6 months.
3. Participants with a history of catastrophic antiphospholipid syndrome are excluded. This includes Participants with a serious thrombotic event (e.g. pulmonary embolism, stroke, deep vein thrombosis) or unexplained pregnancy loss within 1 year before the screening visit or history of 3 or more unexplained consecutive pregnancy losses. Participants with antiphospholipid antibody syndrome on stable anticoagulant therapy at an effective dose are allowed.
4. Participants with active or unstable lupus neuropsychiatric manifestations, including but not limited to any condition defined by BILAG A criteria are excluded, with the exception of participants with mononeuritis multiplex and polyneuropathy, who are allowed.
5. Drug-induced SLE.
6. Participant has a chronic hepatitis B virus (HBV) infection, as defined by positive HBV surface antigen (HBsAg) at screening and detectable HBV core antibody (HBcAb).
7. Participant has chronic hepatitis C virus (HCV) infection, as defined by positive HCV antibody (Ab) at screening and detectable HCV viremia. Participants with positive HCV Ab must undergo reflex HCV ribonucleic acid (RNA) testing, and Participants with HCV RNA positivity will be excluded. Participants with positive HCV Ab and negative HCV RNA are eligible.
8. Participant has a history of or a current immunosuppressive condition or a history of opportunistic infections (e.g. human immunodeficiency virus [HIV] infection, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis, herpes simplex, herpes zoster).
9. Participant testing positive for severe acute respiratory syndrome coronavirus disease 2 (SARS-CoV-2) infection, even if fully vaccinated against SARS-CoV-2, as detected by rapid antigen testing and/or revert transcription polymerase chain reaction (RT-PCR), test at screening and/or baseline (Day 1). Participant presenting any signs or symptoms suggestive of SARS-CoV-2 infection, as detected at screening or baseline following careful physical examination (e.g. cough, fever, headaches, fatigue, dyspnoea, myalgia, anosmia, dysgeusia, anorexia, sore throat), should undergo testing even if fully vaccinated against SARS-CoV-2, as per locally applicable standard diagnostic criteria to diagnose SARS-CoV-2 infection and excluded if positive.
10. Participant meets 1 of the following tuberculosis (TB) criteria at screening:

    * A history of active or currently active TB (regardless of treatment).
    * A positive QuantiFERON®-TB Gold Plus In-tube test at screening unless the investigator assesses this is due to a documented history of adequately treated latent TB infection.

    Note: If the test result is indeterminate, it may be repeated once; if indeterminate or positive on retest, Participant is not eligible.
11. Participant with poorly controlled chronic cardiac, pulmonary, or renal disease.
12. Participant has at screening, presence of severe renal impairment (defined as estimated glomerular filtration rate [eGFR] <30 mL/minute/1.73 m2, using the Chronic Kidney Disease Epidemiology equation).
13. Prior exposure to tyrosine kinase 2 (TYK2) inhibitors.
14. Female participant is pregnant or breast feeding or intending to become pregnant or breastfeed during the study.
15. Participant has taken any prohibited therapies within the defined washout periods before screening, and during screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieved the SLE Responder Index (SRI)-4 Response at Week 32 | Week 32

SECONDARY OUTCOMES:
Percentage of Participants who Achieved the SRI-4 Response at Week 48 | Week 48
Percentage of Participants who Achieved the British Isles Lupus Assessment Group (BILAG)-Based Composite Lupus Assessment (BICLA) Response at Week 32 and Week 48 | Week 32, Week 48
Percentage of Participants with >=50% Reduction in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) score at Week 32 and Week 48 | Week 32, Week 48
Percentage of Participants who achieve Lupus Low Disease Activity State (LLDAS) at Week 32 and Week 48 | Week 32, Week 48
Change from Baseline in the 28-joint Count for Tender joints at Week 32 and Week 48 | Baseline, Week 32 and Week 48
Change from Baseline in the 28-joint Count for Swollen joints at Week 32 and Week 48 | Baseline, Week 32 and Week 48
Change from Baseline in the 28-joint Count for Tender + Swollen (active) joints at Week 32 and Week 48 | Baseline, Week 32 and Week 48
Number of Participants with Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs leading to treatment discontinuation | From the start of first dose till 30 days after the last dose (up to 52 weeks)
Pharmacokinetics (PK) of GLPG3667: Estimated Maximum Plasma Concentration (Cmax) | Predose every 4 weeks from Week 2 to Week 32 and 0.5hours (h)-2h , 2h-4h , 4h-6h postdose at Week 4, Predose every 8 weeks from Week 32 to Week 48
PK of GLPG3667: Estimated Area Under the Concentration Time Curve (AUC) at Steady State | Predose every 4 weeks from Week 2 to Week 32 and 0.5-2h , 2h-4h , 4h-6h postdose at Week 4, Predose every 8 weeks from Week 32 to Week 48
PK of GLPG3667: Estimated Trough Concentration (Ctrough) at Steady State | Predose every 4 weeks from Week 2 to Week 32 and 0.5-2h , 2h-4h , 4h-6h postdose at Week 4, Predose every 8 weeks from Week 32 to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (84):
- United States (22):
  - University of Arizona College of Medicine - Tucson, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - Desert Medical Advances, Rancho Mirage, California
  - Millennium Clinical Trials, Simi Valley, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Upland Rheumatology Center, Upland, California
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - Omega Research DeBary, DeBary, Florida
  - Alloy Clinical Research, LLC, Kissimmee, Florida
  - San Marcus Research Clinic, Miami, Florida
  - Advanced Pharma - Miami, Miami, Florida
  - Professional Research Center, Miami, Florida
  - Integral Rheumatology & Immunology Specialists, Plantation, Florida
  - Alliance Clinical Research of Tampa, Tampa, Florida
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - DJL Clinical Research, Charlotte, North Carolina
  - Lynn Institute of Tulsa, Tulsa, Oklahoma
  - New Phase Research & Development, Knoxville, Tennessee
  - Office of Ramesh C. Gupta MD / Shelby Research LLC - Tennessee, Memphis, Tennessee
  - Care and Cure Clinic, Houston, Texas
  - Southwest Arthritis, Mesquite, Texas
  - Sun Research Institute, San Antonio, Texas
- Argentina (10):
  - Clinica Adventista Belgrano, Belgrano
  - Maffei Centro Medico, Buenos Aires
  - Fundación Respirar - Consultorios Médicos Dr. Doreski, Buenos Aires
  - Fundación Respirar Consultorio Médico Dr. Mariana Rivera, Buenos Aires
  - Investigaciones Reumatológicas y Osteológicas, Caba
  - Clínica Privada Vélez Sarsfield, Córdoba
  - Hospital Italiano La Plata, La Plata
  - Instituto de Reumatología, Mendoza
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes
  - Centro Medico Privado de Reumatología, San Miguel de Tucumán
- Bulgaria (3):
  - Medical Center Artmed, Plovdiv
  - Excelsior Medical Center, Sofia
  - Diagnostic Consultative Center Aleksandrovska, Sofia
- Chile (6):
  - Centro de Estudios Clínicos G y C, Providencia
  - Centros de Estudios Reumatológicos (CER), Providencia
  - Centro Internacional de Estudios Clínicos, Recoleta
  - Prosalud - Centro de Reumatología, Santiago
  - CeCim - Centro de Estudios Clínicos e Investigaciones Médicas, Santiago
  - Oncocentro APYS - Centro de Atención Médica Oncológica Integral, Viña del Mar
- France (3):
  - Hôpital Lapeyronie, Montpellier
  - Hôpital Emile Muller, Mulhouse
  - Hôpital Hautepierre, Strasbourg
- Georgia (5):
  - New Plasma Clinic, Batumi
  - Aversi Clinic - Central Branch, Tbilisi
  - Jerarsi Clinic, Tbilisi
  - Caucasus Medical Center, Tbilisi
  - Clinic Innova LCC, Tbilisi
- Germany (5):
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - LMU Klinikum - Campus Innenstadt, München
  - Praxis Für Rheumatologie, Gastroenterologie Und Innere Medizin, München
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
- Hungary (3):
  - Qualiclinic Egeszsegugyi Szolgaltato es Kutatasszervezo, Budapest
  - Békés Megyei Központi Kórház - Pándy Kálmán Tagkórház, Gyula
  - Vital Medical Center - Reumatológia, Veszprém
- Peru (7):
  - Clínica San Juan de Dios, Cayma
  - ACQ Medic S.A.C., Jesús María
  - Hospital Militar Central Coronel Luis Arias Schreiber, Jesús María
  - Clínica Monterrico, Lima
  - Instituto Peruano Del Hueso Y La Articulacion, San Isidro
  - Clínica Anglo Americana - Sede San Isidro, San Isidro
  - Hospital Maria Auxiliadora, San Juán de Miraflores
- Poland (10):
  - Niepubliczny Zakład Opieki Zdrowotnej Bif-Med S.C., Bytom
  - Centrum Medyczne Plejady, Krakow
  - Poradnie specjalistyczne REUMED Wallenroda, Lublin
  - AES - Synexus - Poznań, Poznan
  - Prywatna Praktyka Lekarska Prof. Dr Hab. Med. Paweł Hrycaj, Poznan
  - Trialmed CRS - Warszawa, Warsaw
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. prof. dr hab. med. Eleonory Reicher, Warsaw
  - Klinika Reuma Park sp. z o.o. sp.k - Centrum Medyczne Reuma Park, Warsaw
  - AES - Synexus - Wrocław, Wroclaw
  - FutureMeds - Wroclaw, Wroclaw
- Puerto Rico (2):
  - Latin Clinical Trial Center, San Juan
  - GCM Medical Group, San Juan
- Spain (8):
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Málaga - Hospital General, Málaga
  - Hospital de Mérida, Mérida
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Araba, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mammoliti O, Martina S, Claes P, Coti G, Blanque R, Jagerschmidt C, Shoji K, Borgonovi M, De Vos S, Marsais F, Oste L, Quinton E, Lopez-Ramos M, Amantini D, Brys R, Jimenez JM, Galien R, van der Plas S. Discovery of GLPG3667, a Selective ATP Competitive Tyrosine Kinase 2 Inhibitor for the Treatment of Autoimmune Diseases. J Med Chem. 2024 Jun 13;67(11):8545-8568. doi: 10.1021/acs.jmedchem.4c00769. Epub 2024 May 28. PMID 38805213